CLINICAL TRIAL: NCT01480310
Title: A Phase Ia, Single-Center, Randomized, Placebo-Controlled, Double-Blind, Single Ascending-Dose Study to Investigate the Safety, Pharmacokinetics, and Immunogenicity of Subcutaneous MCAF5352A in Healthy Volunteers
Brief Title: Study to Investigate the Safety, Pharmacokinetics, and Immunogenicity of Subcutaneous MCAF5352A in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: GA27909
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental)
  Interventions: Drug: MCAF5352A
- B (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MCAF5352A — may receive up to 3 subcutaneous doses of MCAF5352A
  Arms: A
Drug: Placebo — may receive up to 3 subcutaneous doses of placebo
  Arms: B

SUMMARY:
This is a Phase Ia, randomized, double-blind, placebo-controlled, single ascending dose (SAD) study in male and female healthy volunteers, aged 18-55 years, enrolled at a single study site in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Total body weight between 45 and 110 kg
* Vital signs within the following ranges: oral body temperature of 35°C to 37.5°C, systolic blood pressure of 90 to 140 mmHg, diastolic blood pressure of 50 to 90 mmHg, and pulse rate of 45 to 100 bpm
* Laboratory test parameters within normal reference ranges of the safety laboratory
* Female subjects: Willing to use two effective methods of contraception from screening to a minimum of 4 months after the last dose of study drug. Reliable forms of contraception include oral hormonal contraceptives, patch hormonal contraceptives, vaginal ring, intrauterine device, physical double-barrier methods, surgical hysterectomy, or vasectomy by male partner.

Exclusion Criteria:

* Pregnant or lactating women
* Administration of a live, attenuated vaccine within 30 days before Day 1 or anticipation that such a live attenuated vaccine will be required within 100 days of Day 1
* Subjects may receive influenza vaccination only during influenza season (approximately October to March). Subjects must not receive live attenuated influenza vaccine within 30 days prior to Day 1 or at any time during the study.
* Any major illness within 30 days prior to Day 1
* Clinically significant illness requiring treatment within 14 days prior to Day 1
* History of clinically significant ECG abnormalities or a known family history of cardiac conduction system disease
* Positive test results indicating current or past infection with human immunodeficiency virus (HIV-1 or 2), hepatitis B virus (hepatitis B surface antigen [HBsAg], hepatitis B core antibody [anti-HBc]), or hepatitis C virus (HCV)
* Positive screening test for latent mycobacterial infection within the 2 months preceding Day 1 without evidence of a completed course of anti-tubercular therapy or previous BCG vaccination
* History of significant chronic or recurrent infections
* History of clinically significant drug allergy and/or a known hypersensitivity to protein therapeutics or formulation components or a related drug
* History of alcohol or drug abuse within 12 months prior to Day 1, or evidence of such abuse as indicated by the specific screening laboratory tests results, or alcohol consumption of more than 14 units of alcohol per week
* Positive breathalyzer for alcohol or urine screen results for drugs of abuse, or prescription medications
* Subjects who have previously received the study drug
* Participation in a clinical trial within 4 weeks before Day 1 or use of any experimental or biologic therapy within the 12 weeks prior to Day 1 or within 5 half-lives of the product, whichever is greater
* Use of prescription drugs within 14 days prior to Day 1 or during the study, except for hormonal contraceptives or hormone replacement therapy
* Use of over-the-counter (OTC) medication within 7 days prior to Day 1 or during the study. Medications such as acetaminophen and ibuprofen and routinely-taken dietary supplements, including vitamins and herbal supplements are allowed at the discretion of the investigator and provided that the medication in question has no discernible impact on the study.
* Donation of plasma within 7 days prior to Day 1. Donation or loss of blood of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to Day 1.
* Lack of peripheral venous access
* Known history of mental illness

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | up to approximately 100 days

SECONDARY OUTCOMES:
Pharmacokinetic: maximum serum concentration (Cmax) | up to approximately 100 days
Pharmacokinetic: time to maximum serum concentration (tmax) | up to approximately 100 days
Pharmacokinetic: apparent clearance (CL/F) | up to approximately 100 days
Pharmacokinetic: Terminal half-life (t½) | up to approximately 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Québec, Quebec, Canada